CLINICAL TRIAL: NCT06514170
Title: Assessment of Gastrointestinal Dysfunction Through GIDS Scale and Intestinal Damage Biomarkers in Critically Ill Patients Undergoing Aortic Surgery and Its Association With Clinical Outcomes.
Brief Title: Gastrointestinal Dysfunction in Aortic Surgery Patients
Status: Recruiting | Type: Observational
Sponsor: Instituto Nacional de Cardiologia Ignacio Chavez (Other)
Collaborators: Instituto Nacional de Enfermedades Respiratorias (Other Government); National Polytechnic Institute, Mexico (Other)
Responsible Party: Principal Investigator, Gustavo Rojas Velasco, Head of the Cardiovascular Intensive Care Unit, Instituto Nacional de Cardiologia Ignacio Chavez
Other Study IDs: 24-1427
Record Dates: First submitted 2024-07-09; First posted 2024-07-23 (Actual); Last update posted 2024-07-24 (Actual); Status verified 2024-07

CONDITIONS: Aortic Aneurysm; Gastrointestinal Dysfunction; Aortic Diseases; Enteral Feeding Intolerance; Surgical Complication
Keywords: Gastrointestinal dysfunction; Aortic diseases; Aorta surgery
MeSH Terms: conditions — Aortic Aneurysm; Aortic Diseases

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood samples will be collected, which will then be processed to obtain plasma for the determination of citrulline and I-FABP biomarkers on days 1, 3, and 5 of ICU stay.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: No intervention — No intervention

SUMMARY:
The goal of this observational study is to determine the association of gastrointestinal dysfunction through the Gastrointestinal Dysfunction Scale (GIDS) tool and serum concentrations of citrulline and Intestinal fatty-acid binding protein (I-FABP) with primary [calories received, protein received, parenteral nutrition requirement and 28-day mortality in the intensive care unit (ICU)] and secondary (development of pneumonia, surgical and cardiovascular complications in the ICU, length of hospital and ICU stay, duration of mechanical ventilation) clinical outcomes in critically ill patients undergoing aortic surgery.

DETAILED DESCRIPTION:
The treatment of choice for various cardiovascular diseases often involves cardiac surgery, including aortic surgery, which is performed to correct conditions related to this major vessel, such as aneurysms, stenosis, aortic dissections, as well as issues affecting the aortic valve. With the increasing prevalence of non-communicable chronic diseases, a 46% increase in demand for cardiac surgeries is projected by 2025. The post-surgical period, commonly in the intensive care unit (ICU), increases the risk of complications, especially in patients with pre-existing risk factors. In this regard, gastrointestinal (GI) dysfunction affects up to 63% of patients, being associated with complications and a mortality rate of 55% to 60%. Early detection of GI dysfunction allows for the implementation of management strategies. Additionally, the administration of appropriate nutritional therapy is essential for recovery, and GI dysfunction may limit nutrient absorption. Inadequate caloric intake has been linked to increased morbidity and mortality. Tools such as GIDS (Gastrointestinal Dysfunction Scale) and biomarkers like citrulline and I-FABP enable early evaluation of GI function, advancing monitoring and management. Identifying changes before serious complications arise allows for early and personalized interventions. Early detection not only prevents complications and improves quality of life but may also reduce mortality. This research project aims to address these gaps by early assessing GI dysfunction in post-aortic surgery patients. Utilizing the GIDS tool and biomarkers such as citrulline and I-FABP, the goal is to identify GI dysfunction early and its impact on nutrition administration.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older.
* Patients after surgical interventions (elective or urgency) on the aorta with cardiopulmonary bypass.
* Invasive mechanical ventilation expected to be required more than 48 hours.
* Signed informed consent.

Exclusion Criteria:

* Patients under mechanical ventilation with pre-existing gastrointestinal issues.
* Diagnosis of adult congenital heart disease.
* Ongoing pregnancy or lactation period.
* Simultaneous participation in another clinical study involving experimental therapy.
* Presence of chronic intestinal disease.
* Previous gastrointestinal conditions detected during nutritional screening.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients following aortic surgery necessitating invasive mechanical ventilation and an intensive care unit stay of ≥ 48 hours.
Sampling Method: Probability Sample
Enrollment: 114 (Estimated)
Dates: Start 2024-07-23 (Actual); Primary Completion 2026-04 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Calories delivered daily enterally and/or parenterally | Day 0 to day 7
  Percentage representation of prescribed calories delivered daily via enteral and/or parenteral routes.
Protein delivered daily enterally and/or parenterally | Day 0 to day 7
  Daily administration of protein (in grams) through enteral and/or parenteral routes.

SECONDARY OUTCOMES:
Incidence rate of hospital-acquired infections | 7 days
  Infections acquired in the hospital consist of ventilator-associated pneumonia, bloodstream infections, and infections related to urinary catheters
Percentage of repeated operations | 90 days
  This outcome measures the percentage of patients who undergo one or more additional surgical operations related to the same condition after the initial surgery. The percentage is calculated by dividing the number of patients who require a repeat operation by the total number of patients who underwent the initial operation, multiplied by 100 to get the percentage.
ICU readmission rate | 90 days
  Occurrences of patients being readmitted to the ICU from within the hospital.
ICU length of stay | 90 days
  Duration of time (days) in the ICU
Duration of mechanical ventilation | 90 days
  Length of time (days) on mechanical ventilation (including still on mechanical ventilation at time of discharge)
Hospital length of stay | 90 days
  Duration of time (days) in the hospital
Parenteral nutrition requirement | Day 0 to day 7
  Parenteral nutrition requirement
28-day mortality in the ICU | 28 days
  Is the patient alive or deceased 28 days post admission.

CONTACTS AND LOCATIONS:
Overall Officials: Gustavo Rojas Velasco, MD, Principal Investigator — Head of the Cardiovascular Intensive Care Unit
Locations (1):
- Instituto Nacional de Cardiología Ignacio Chávez, Mexico City, Tlalpan, Mexico

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Stoppe C, Spillner J, Rossaint R, Coburn M, Schalte G, Wildenhues A, Marx G, Rex S. Selenium blood concentrations in patients undergoing elective cardiac surgery and receiving perioperative sodium selenite. Nutrition. 2013 Jan;29(1):158-65. doi: 10.1016/j.nut.2012.05.013. Epub 2012 Sep 23. PMID 23010420
- [Background] Reintam Blaser A, Preiser JC, Fruhwald S, Wilmer A, Wernerman J, Benstoem C, Casaer MP, Starkopf J, van Zanten A, Rooyackers O, Jakob SM, Loudet CI, Bear DE, Elke G, Kott M, Lautenschlager I, Schaper J, Gunst J, Stoppe C, Nobile L, Fuhrmann V, Berger MM, Oudemans-van Straaten HM, Arabi YM, Deane AM; Working Group on Gastrointestinal Function within the Section of Metabolism, Endocrinology and Nutrition (MEN Section) of ESICM. Gastrointestinal dysfunction in the critically ill: a systematic scoping review and research agenda proposed by the Section of Metabolism, Endocrinology and Nutrition of the European Society of Intensive Care Medicine. Crit Care. 2020 May 15;24(1):224. doi: 10.1186/s13054-020-02889-4. PMID 32414423
- [Background] van Zanten AR. Nutrition barriers in abdominal aortic surgery: a multimodal approach for gastrointestinal dysfunction. JPEN J Parenter Enteral Nutr. 2013 Mar;37(2):172-7. doi: 10.1177/0148607112464499. Epub 2012 Oct 24. No abstract available. PMID 23100540
- [Background] Reintam Blaser A, Padar M, Mandul M, Elke G, Engel C, Fischer K, Giabicani M, Gold T, Hess B, Hiesmayr M, Jakob SM, Loudet CI, Meesters DM, Mongkolpun W, Paugam-Burtz C, Poeze M, Preiser JC, Renberg M, Rooijackers O, Tamme K, Wernerman J, Starkopf J. Development of the Gastrointestinal Dysfunction Score (GIDS) for critically ill patients - A prospective multicenter observational study (iSOFA study). Clin Nutr. 2021 Aug;40(8):4932-4940. doi: 10.1016/j.clnu.2021.07.015. Epub 2021 Jul 18. PMID 34358839
- [Background] Liu X, Wang Q, Yang D, Fu M, Yang M, Bi Y, Wang C, Song X. Association between Gastrointestinal Dysfunction Score (GIDS) and disease severity and prognosis in critically ill patients: A prospective, observational study. Clin Nutr. 2023 May;42(5):700-705. doi: 10.1016/j.clnu.2023.03.004. Epub 2023 Mar 7. PMID 36958226